CLINICAL TRIAL: NCT06680622
Title: Bemarituzumab in Patients With FGFR2b-positive Advanced or Metastatic Adenocarcinoma of the Stomach or Gastroesophageal Junction, Who Failed at Least One Prior Line of Palliative Chemotherapy - The IKF-AIO Phase IIa BEMARA Trial
Brief Title: Bemarituzumab in FGFR2b+ Patients With Advanced or Metastatic Adenocarcinoma of the Stomach or Gastroesophageal Junction, Who Failed at Least One Prior Line of Palliative Chemotherapy
Status: Active, not recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Institut für Klinische Krebsforschung IKF GmbH at Krankenhaus Nordwest (Other)
Collaborators: Amgen (Industry); Johannes Gutenberg University Mainz (Other); Technical University of Munich (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: BEMARA; 2024-512484-31-00 (EU CTIS Number)
Record Dates: First submitted 2024-11-01; First posted 2024-11-08 (Actual); Last update posted 2026-01-07 (Actual); Status verified 2026-01

CONDITIONS: Metastatic Gastro-esophageal Adenocarcinoma
Keywords: BEMARA; FGFR2b; adenocarcinoma of the stomach or gastroesophageal junction
MeSH Terms: interventions — bemarituzumab; Paclitaxel; Ramucirumab; Irinotecan; Trifluridine; tipiracil

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Cohort 1 (Experimental): bemarituzumab plus SOC treatment with irinotecan
  Interventions: Drug: bemarituzumab, irinotecan
- Cohort 2 (Experimental): bemarituzumab plus SOC treatment with paclitaxel plus ramucirumab
  Interventions: Drug: bemarituzumab, paclitaxel, ramucirumab
- Cohort 3 (Experimental): bemarituzumab plus SOC treatment with trifluridine/tipiracil
  Interventions: Drug: bemarituzumab, trifluridine/tipiracil

INTERVENTIONS:
Drug: bemarituzumab, paclitaxel, ramucirumab — Cohort 2 will receive bemarituzumab plus SOC treatment with paclitaxel and ramucirumab
  Arms: Cohort 2
Drug: bemarituzumab, irinotecan — Cohort 1 will receive bemarituzumab plus SOC treatment with irinotecan
  Arms: Cohort 1
Drug: bemarituzumab, trifluridine/tipiracil — Cohort 3 will receive bemarituzumab plus SOC treatment with trifluridine/tipiracil
  Arms: Cohort 3

SUMMARY:
The goal of this clinical trial is to evaluate if bemarituzumab in combination with different standard of care chemotherapies enhance tumor response in patients with FGFR2b-positive advanced or metastatic adenocarcinoma of the stomach or gastroesophageal junction. The main questions are:

How do patients respond to these treatments? How is the overall and the progression-free survival rate with these treatments? How is the disease control rate with these treatments? How long is the duration of response and disease stabilization with these treatments? How is the safety with these treatments? How is the quality of life with these treatments?

Patients will be allocated to one of three possible treatment cohorts according to investigator's decision and current standard of care:

Bemarituzumab with cohort 1: irinotecan cohort 2: paclitaxel plus ramucirumab cohort 3: trifluridine/tipiracil

ELIGIBILITY:
Inclusion Criteria:

1. Patient provide signed informed consent form.
2. Patient is ≥ 18 years at the time of given informed consent.
3. Patient has been diagnosed with histologically proven advanced or metastatic adenocarcinoma of the stomach or of the gastroesophageal junction, which is not amenable to potentially curative resection. Primary tumor locations will be classified following AJCC/UICC 8th ed.
4. Patient has measurable disease or non-measurable, but evaluable disease, according to RECIST v1.1
5. Patient received at least one previous line of treatment, which includes a fluoropyrimidine and a platinum, in the advanced setting or the patient has been intolerable or ineligible to fluoropyrimidine and/or platinum. Neoadjuvant/adjuvant treatment is not counted unless progression occurs <6 months after completion of the treatment. In these cases, neoadjuvant/adjuvant treatment is counted as one line of therapy.

   Note: patient allocation to cohort 3 only if patient received at least two previous lines of treatment.
6. Tumor material (archival and/or fresh) is available for centrally FGFR2b testing performed by IHC.

   • FGFR2b-selected population using 2+/3+ definition in ≥ 10% tumor cells.
7. Patients with HER2/neu-positive tumors are eligible if they received prior HER2/neu-targeted therapy.
8. Patient has an ECOG performance status ≤ 1.
9. Patient has a life expectancy > 12 weeks.
10. Patient has adequate hematological, hepatic and renal function.

    1. Absolute number of neutrophils (ANC) ≥ 1.5 x 109/L
    2. Platelets ≥ 100 x 109/L
    3. Hemoglobin ≥ 9 g/dL (5.58 mmol/L), without transfusion support within 7 days before the first dose of study treatment
    4. Total bilirubin ≤ 1.5 times the upper limit of normal (ULN) (or < 2 x ULN in case of liver involvement or Gilbert's disease)
    5. AST (SGOT) and ALT (SGPT) ≤ 2.5 x ULN without existing liver metastases, or ≤ 5 x ULN in the presence of liver metastases; AP ≤ 5 x ULN
    6. Serum creatinine ≤ 1.5 x ULN or creatinine clearance (measured by 24 h urine) ≥ 50 mL/min (i.e., if serum creatinine level is > 1.5 x ULN, then a 24-hour urine test must be performed to check the creatinine clearance to be determined).
11. Adequate coagulation function as defined by International Normalized Ratio (INR) ≤ 1.5, and a partial thromboplastin time (PTT) ≤ 5 seconds above the ULN (unless receiving anticoagulation therapy).
12. Female patients of childbearing potential, as defined in Section 5.1.7, or male patients with female partners of childbearing potential must agree to remain abstinent (refrain from heterosexual intercourse) or use contraceptive methods that result in a failure rate of <1% (see Section 5.1.7) per year during the treatment period and for at least 6 months after the last trial treatment. Male patients must agree not to donate sperm within the same period. Male patients with a pregnant partner must agree to remain abstinent or to use a condom for the duration of the pregnancy. Female patients of child-bearing potential must have a negative pregnancy test within the last 7 days prior to the start of trial therapy.
13. Patient is willing and able to comply with the protocol (including contraceptive measures) for the duration of the study including undergoing treatment and scheduled visits and examinations including follow up

Exclusion Criteria:

1. Patient received prior treatment any selective inhibitor of the FGF-FGFR pathway or participated in a study that randomized to FGFR-targeted therapy/placebo.
2. Patient has known allergic / hypersensitive reactions to at least one of the treatment components
3. Contraindication for standard of care (SOC) treatment regimen chosen by investigator (irinotecan, paclitaxel plus ramucirumab or trifluridine/tipiracil) according to specific product information or clinical standards
4. Patient has known presence of tumors other than adenocarcinomas (e.g., leiomyosarcoma, lymphoma) or a secondary tumor other than squamous or basal cell carcinomas of the skin or in situ carcinomas of the cervix which have been effectively treated. The sponsor decides to include patients who have received curative treatment and have been disease-free for at least 5 years.
5. Patient has squamous/ adenosquamous cell carcinoma of the stomach or gastroesophageal junction.
6. Patient receives simultaneous, ongoing, systemic immunotherapy, chemotherapy, hormone therapy or investigational treatment not described in the study protocol.
7. Patient receives current treatment with any anti-cancer therapy or major surgery ≤ 2 weeks prior to study treatment start unless rapidly progressing disease is measured.
8. Patient receives simultaneous treatment with a different anti-cancer therapy (including investigational treatments) other than that provided for in the trial (excluding palliative radiotherapy for symptom control).
9. Patient has known untreated or symptomatic CNS or leptomeningeal metastases. Subjects with asymptomatic CNS metastases are eligible if clinically stable for ≥ 4 weeks and require no intervention (including use of corticosteroids). Subjects with treated brain metastases are eligible provided the following criteria are met:

   1. Definitive therapy was completed at least 2 weeks prior to the first planned dose of trial treatment (stereotactic radiosurgery at least 7 days prior to first planned dose of study treatment)
   2. At least 7 days prior to first dose of trial treatment: any CNS disease is clinically stable, subject is off steroids for CNS disease (unless steroids are indicated for a reason unrelated to CNS disease), and subject is off or on stable doses of anti-epileptic drugs
10. Patient has impaired cardiac function or clinically significant cardiac disease including unstable angina within 6 months before the first dose of study treatment, acute myocardial infarction < 6 months prior to the first dose of study treatment, New York Heart Association (NYHA) class II-IV congestive heart failure, uncontrolled hypertension (defined as an average systolic blood pressure > 160 mmHg or diastolic > 100 mmHg despite optimal treatment, uncontrolled cardiac arrhythmias requiring antiarrhythmic therapy other than beta blockers or digoxin, active coronary artery disease or corrected QT interval (QTc) ≥ 470
11. Patient has evidence of or any ongoing ophthalmological disorders.

    1. History of systemic disease or ophthalmologic disorders requiring chronic use of ophthalmic steroids
    2. Evidence of any ongoing ophthalmologic abnormalities or symptoms that are acute (within 4 weeks) or are actively progressing
    3. Unwillingness to avoid use of contact lenses during study treatment and for ≥ 100 days after the end of treatment
    4. Recent (within 6 months) corneal surgery or ophthalmic laser treatment or recent (within 6 months) history of, or evidence of corneal defects, corneal ulcerations, keratitis, or keratoconus, or other known abnormalities of the cornea that may pose an increased risk of developing a corneal ulcer
12. Patient has a serious infection requiring oral or IV antibiotics within 14 days prior to trial enrollment.
13. Patient has an acute or chronic infection with human deficiency virus (HIV), or an acute infection with hepatitis B or C virus (HBV, HCV). Exception: Subjects with hepatitis B surface antigen or core antibodies who achieve a sustained virologic response with antiviral therapy directed against hepatitis B and subjects with hepatitis C, who achieve a sustained virologic response following antiviral therapy are permitted.
14. Patient experienced severe, life-threatening, or recurrent (Grade 2 or higher) immune-mediated adverse events (AEs) or infusion-related reactions including those that led to permanent discontinuation while on treatment with immune-oncology agents
15. Patient received prior immunosuppressive therapy: immunosuppressive doses of systemic medications of > 10 mg/day of prednisone or equivalent must be discontinued ≥ 2 weeks before the first dose of study treatment. Short courses of high dose corticosteroids and/or continuous low dose of prednisone (< 10 mg/day) are permitted. In addition, inhaled, intranasal, intraocular, and/or joint injections of corticosteroids are allowed
16. Patient has evidence of any other serious concomitant or medical condition that, in the opinion of the investigator, presents a high risk of complications to the patient or reduces the likelihood of clinical effect.
17. Female patient is pregnant or breast feeding or planning to become pregnant within and up to 4 months after end of treatment (if enrolled to Cohort 1) or up to 6 months after the end of treatment (if enrolled to Cohort 2 or 3).

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 126 (Estimated)
Dates: Start 2025-03-03 (Actual); Primary Completion 2027-09 (Estimated); Study Completion 2028-03 (Estimated)

PRIMARY OUTCOMES:
Objective response rate (ORR) | from date of enrollment to date of last response acc. to RECIST v1.1 or death due to any cause, through study completion, up to 33 months
  Objective response rate (ORR), defined as proportion of subjects with a complete response (CR) or partial response (PR) acc. to RECIST v1.1, for each cohort (cohort 1 - bemarituzumab plus irinotecan, cohort 2 - bemarituzumab plus paclitaxel and ramucirumab, cohort 3 - bemarituzumab plus trifluridine/tipiracil).

SECONDARY OUTCOMES:
Progression-free survival (PFS) | from date of enrollment to date of progression acc. to RECIST v1.1 or death due to any cause, through study completion, up to 33 months
  Progression-free survival (PFS)
Overall survival (OS) | time from date of enrollment to date of death due to any cause, through study completion, up to 33 months
  Overall survival (OS)
Disease control rate (DCR) | time from date of enrollment to date of last tumor assessment acc. to RECIST 1.1 or death due to any cause, through study completion, up to 33 months
  proportion of subjects with CR, PR or stable disease (SD) according to RECIST v1.1
Duration of response (DoR) | time from response initiation (when either CR or PR is first determined) to date of progression or death to any cause, through study completion, up to 33 months
  Duration of response (DoR)
Disease stabilization | time from the first assessment of CR or PR or SD until the date of progression or death to any cause, through study completion, up to 33 months
  Duration of disease stabilization
Quality of Life (QoL) with EORTC QLQ C30 | time from baseline questionnaire to last filled questionnaire in follow up or until progression or death of any cause, through study completion, up to 33 months
  Assessment of quality of life using EORTC QLQ C30 questionnaires during treatment
Quality of Life (QoL) with EQ-5D-5L | time from baseline questionnaire to last filled questionnaire in follow up or until progression or death of any cause, through study completion, up to 33 months
  Assessment of quality of life using EQ-5D-5L visual analogue scale (VAS) score
Quality of Life (QoL) with HADS | time from baseline questionnaire to last filled questionnaire in follow up or until progression or death of any cause, through study completion, up to 33 months
  Assessment anxiety/depression and satisfaction using HADS during treatment

CONTACTS AND LOCATIONS:
Overall Officials: Sylvie Lorenzen, Prof. Dr., Principal Investigator — Klinikum München rechts der Isar der Technischen Universität München; Salah Eddin Al-Batran, Prof. Dr., Study Chair — Frankfurter Institut für Klinische Krebsforschung IKF GmbH
Locations (35):
- Germany (35):
  - Uniklinik RWTH Aachen, Aachen
  - Klinikum St. Marien, Amberg
  - Universitätsklinikum Augsburg, Augsburg
  - Helios Klinikum Bad Saarow, Bad Saarow
  - Klinikum Neukölln Vivantes Netzwerk für Gesundheit GmbH Klinlinik für Innere Medizin - Hämatologie und Onkologie, Berlin
  - Charité - Universitätsmedizin Berlin Medizinische Klinik mit Schwerpunkt Hämatologie, Onkologie und Tumorimmunologie (CVK), Berlin
  - VIVANTES Berlin Friedrichshain, Berlin
  - Klinikum Bielefeld gem. GmbH Klinik für Hämatologie, Onkologie und Palliativmedizin, Bielefeld
  - Klinikum Chemnitz, Chemnitz
  - St.-Johannes-Hospital, Dortmund
  - Gemeinschaftspraxis Hämatologie-Onkologie, Dresden
  - Universitätsklinikum Düsseldorf Klinik für Gastroenterologie, Hepatologie und Infektiologie Gastroonkologische Studienzentrale, Düsseldorf
  - Kliniken Essen-Mitte, Essen
  - Krankenhaus Nordwest GmbH Institut für Klinisch-Onkologische Forschung (IKF), Frankfurt
  - Universitätsklinikum Gießen und Marburg GmbH Standort Gießen Medizinische Klinik IV; Organonkologie Studienzentrale, Giessen
  - Universität Göttingen, Göttingen
  - Onkodoc Gütersloh, Gütersloh
  - Hämatologisch-Onkologische Praxis Eppendorf (hope) Norddeutsches Studienzentrum für Innovative Onkologie, Hamburg
  - MH Hannover, Hanover
  - Universitätsklinikum Heidelberg Nationales Centrum für Tumorerkrankungen (NCT Heidelberg), Heidelberg
  - St. Anna Hospital Herne, Herne
  - Universitätsklinikum Jena, Jena
  - Universitätsklinikum Schleswig-Holstein, Kiel
  - Medizinisches Versorgungszentrum Landshut, Landshut
  - Universitäres Krebszentrum Leipzig (UCCL), Leipzig
  - Klinikum Magdeburg, Magdeburg
  - Universitätsmedizin Mainz I. Medizinische Klinik und Poliklinik, Mainz
  - Klinikum rechts der Isar der technischen Univeristät München Medizinische Klinik und Poliklinik III Hämatologie und Onkologie, München
  - Klinikum der Universität München Med. Klinik und Poliklinik III AG Onkologie, München
  - Klinikum München-Bogenhausen, München
  - Universitätsklinikum Regensburg, Regensburg
  - Krankenhaus Barmherzige Brüder Regensburg Klinik für Onkologie und Hämatologie, Regensburg
  - Kreiskliniken Reutlingen gGmbH Klinikum am Steinenberg Reutlingen/Medizinische Klinik I, Reutlingen
  - HELIOS Kliniken Schwerin, Schwerin
  - Klinikum Wolfsburg Medizinische Klinik II, Wolfsburg

IPD SHARING:
Plan to Share IPD: No
No IPD will be shared